CLINICAL TRIAL: NCT04100876
Title: Effect of DNA Methyltransferase 3A-448 G/A and 3B-149 C/T Single Nucleotide Polymorphisms on Global DNA Methylation in Primary Immune Thrombocytopenia
Brief Title: Effect of DNMT SNPs on DNA Methylation in Primary ITP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennat-Allah Abdelnasser Mahmoud Ahmed, Clinical Pathology Department, Assiut University
Other Study IDs: DNA methylation in Primary ITP
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Study will be conducted on DNA samples (available from previous study of AbdelKader et al., 2018) with known DNMT3A -448 G/A and DNMT3B -149C/T genotypes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- primary ITP patients .: 60 primary ITP patients .
  Interventions: Genetic: Global DNA methylation will be quantified in the DNA samples by colorimetry
- healthy subjects .: 30 healthy age and sex matched control subjects .
  Interventions: Genetic: Global DNA methylation will be quantified in the DNA samples by colorimetry

INTERVENTIONS:
Genetic: Global DNA methylation will be quantified in the DNA samples by colorimetry — Global DNA methylation will be quantified in the DNA samples by colorimetry

SUMMARY:
* To compare global DNA methylation status between ITP patients and healthy subjects .
* To determine the effect of DNMT3A -448 G/A SNP variant A allele and DNMT3B -149C/T SNP variant T-allele on global DNA methylation in both ITP patients and healthy control subjects.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP), is an immune-mediated acquired disease of adults and children characterized by transient or persistent decrease of the platelet count and, depending upon the degree of thrombocytopenia, increased risk of bleeding (Rodeghiero et al., 2009). International guidelines define thrombocytopenia as a peripheral blood platelet count less than 100 000/uL (Raj, 2017). Platelet count values between 100 000/uL and 150 000/uL are frequently found in apparently healthy people (Adibi et al., 2007) and this threshold reduces the concern over the mild "physiologic" thrombocytopenia associated with pregnancy (Neunert et al., 2011).

Immune thrombocytopenia may be primary or secondary. Primary ITP is a diagnosis of exclusion. Secondary ITP occur due to an underlying diseases/conditions. Causes of secondary ITP include infection (CMV, Helicobacter pylori, HCV, HIV, Varicella zoster), Systemic lupus erythematosus, Antiphospholipid syndrome, Drug-induced, Lymphoproliferative disorders, Post bone marrow transplantation, and Post vaccination (Neunert et al., 2011).

Primary ITP is an acquired autoimmune disease causing both increased platelet destruction and insufficient platelet production. More than one mechanism could contribute to this including autoreactive B lymphocytes, Th1/Tc1 polarization, T-cell-mediated platelet lysis and abnormal circulating Treg cells. Also, DNA methylation may participate in the pathophysiology of ITP (Semple et al., 2010, Wang et al., 2011).

DNA methylation is a heritable, stable, and also reversible way of DNA modification; it can regulate gene expression without changing the nucleotide sequences (Huiyuan et al., 2013). DNA methylation is mediated by DNA methyltransferases (DNMTs). There are five members in DNMT group including DNMT3A and DNMT3B (Okano et al., 1999). DNMT3A and DNMT3B catalyze de novo methylation and it is important in the establishment of DNA methylation patterns within the embryo and during fetal development (Sawalha, 2008).

DNA methylation status takes part in the regulation of immune response, the loss of methylation pattern in immune cells will result in autoimmune disease by inducing aberrant gene expression. ITP is an autoimmune disease with many immune deficiencies with abnormal DNA methylation involved in the disease etiology (Huiyuan et al., 2013). Chen et al., 2011, concluded that aberrant DNA methylation may take part in the pathogenesis of ITP by quantifying the methylcytosine concentration of genomic DNA. They found hypomethylation pattern in CD4 T cells of ITP patients.

DNMT3A, and DNMT3B DNA methyltransferases are encoded by different genes on distinct chromosomes (Sawalha, 2008). There are many single nucleotide polymorphisms (SNPs) in DNMT3A gene which may affect catalytic activity of the DNMT3A enzyme, including -448G/A SNP (Zhao et al., 2012). Twenty-one polymorphisms have been identified in the DNMT3B gene including -149 C/T SNP and -579 G/T SNP (Zhang et al., 2015).

In a previous study in Assiut University Hospital (AbdelKader et al., 2018), the DNMT3A -448 G/A SNP variant A allele was significantly associated with decreased risk of primary ITP, while, DNMT3B -149C/T SNP variant T-allele was significantly associated with nearly double-fold increase in risk of primary ITP. However, the underlying mechanism behind this association was not investigated. Authors recommended to study mRNA expression of DNMT genes, enzymatic activity of DNA methyltransferases, quantification of global methylated DNA, and/or methylation status of methylation-sensitive genes involved in primary ITP pathogenesis to understand this association.

ELIGIBILITY:
Inclusion Criteria:

* . Egyptian patients with isolated thrombocytopenia, no organomegaly or lymphoadenopathy, no constitutional symptoms (bone pains, weight loss, and night sweats) and no history of preceding drug intake (quinine, heparin) .

Exclusion Criteria:

* Conditions/diseases associated with secondary ITP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: : 60 primary ITP patient and 30 healthy age and sex matched control subjects .
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of global DNA methylation status between ITP patients and healthy subjects . | baseline .
  To understand the underlying mechanism behind the association of DNMT3A -448 G/A SNP variant A allele with decreased risk of primary ITP and DNMT3B -149C/T SNP variant T-allele with increased risk of primary ITP which was observed in a previous study in Assiut University Hospital (AbdelKader et al., 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Heba A Abdel-Hafeez, Professor, Study Director — Clinical Pathology Department in Assuit University Hospital